CLINICAL TRIAL: NCT02252783
Title: A Phase II Open-Labeled Study to Evaluate BFPET as a Myocardial Perfusion Imaging Agent for the Evaluation of Coronary Artery Disease
Brief Title: BFPET for Regional Myocardial Perfusion Imaging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fluoropharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BFPET P-02
Record Dates: First submitted 2014-09-25; First posted 2014-09-30 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BFPET (Experimental): BFPET will be administered as a single intravenous injection of up to 2 mCi (74 MBq) at rest and a single intravenous injection of up to 8mCi (296 MBq) following a stress protocol. Total amount not to exceed 10mCi (370 MBq).
  Interventions: Drug: BFPET

INTERVENTIONS:
Drug: BFPET — Sterile study drug will be delivered in individual dosage vials labeled and calibrated to approximately 2 mCi (74MBq) for the rest imaging and up to 8 mCi (296 MBq) for the stress imaging at the time of injection. The drug will be administered intravenously by bolus injection over 10 seconds into a peripheral vein to which access has been secured followed by saline flush.
  Other Names: FTPP FluorophenylTriPhenylPhosphonium

SUMMARY:
BFPET will be evaluated as a diagnostic PET agent for assessing myocardial perfusion in subjects with known or suspected coronary artery disease (CAD) as compared to standard nuclear myocardial perfusion imaging (MPI). The safety of BFPET will be evaluated in known or suspected CAD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to any study related procedures;
* Subjects must be ≥ 21 and ≤ 85 years of age;
* Subjects must have known or suspected CAD documented by ≥2 segments of reversible perfusion abnormalities on a SPECT (MPI)study

Exclusion Criteria

* Any clinically significant acute or unstable physical or psychological disease judged by the investigators based on medical history or screening physical examination;
* Blood pressure over 180/100mmHg
* Acute changes in comparison to most recent ECG;
* Recent (within 3 months) cardiac arrest, unstable angina, cerebro-vascular accident (CVA), CABG or PCI
* Any pacemaker or defibrillator implanted within the last three months;
* Inability to remain in camera for approximately 60 minutes
* Bronchospasm
* Serum creatinine > 2 mg/dL;
* Cancer patients who have received chemotherapy or radiation therapy within the past 60 days.
* Any exposure to any investigational drug(s) or medical device(s) within four (4) weeks prior to imaging study;
* Any physical or psychological disease judged by the investigators to be incompatible with the study, based on medical history or screening physical examination.
* NYHA Class III or IV Congestive heart failure;
* Subject has symptomatic hypotension
* Allergic or intolerant to aminophylline, nitroglycerin or metoprolol
* Allergic or intolerant to regadenoson or any of its excipients
* Prior participants in the study.
* Female subjects only: Positive serum and/or urine pregnancy test or is lactating or the possibility of pregnancy cannot be ruled out prior to dosing.

Females not of child-bearing potential require confirmatory documentation in their medical records or must have a negative pregnancy test within 4 hours prior to receiving the test drug and agree to use an acceptable form of birth control for at least 30 days following BFPET administration.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of BFPET | Up to 30 days
  To evaluate the diagnostic performance of BFPET as a PET agent assessment of myocardial perfusion in known or suspected CAD subjects.

SECONDARY OUTCOMES:
Primary safety endpoints - ECG, physical examinations, vital signs, laboratory and adverse event assessments | Up to 10 days
  Vital signs, ECG, laboratory assessments - up to 24 hours post injection, adverse event assessment at all study visits (7-10 days) post BFPET administration

CONTACTS AND LOCATIONS:
Overall Officials: Georges El Fakhri, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided